CLINICAL TRIAL: NCT00550797
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Crossover Study to Evaluate the Safety and Efficacy of 14-day Inhaled TPI ASM8 in Subjects With Asthma
Brief Title: Study to Evaluate the Safety and Efficacy TPI ASM8 in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Collaborators: i3 Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPI ASM8-205
Record Dates: First submitted 2007-10-26; First posted 2007-10-30 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Allergic Asthma
Keywords: Steroid-naive, non-smokers; Mild to moderate allergic asthmatic adults
MeSH Terms: interventions — TPI ASM8

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No.1 ASM8 (oligonucleotide) (Experimental): TPI ASM8 1mg/mL in phosphate buffered saline (PBS) solution; 1 mg will be administered daily (morning) by inhalation
  Interventions: Biological: TPI ASM8
- Phosphate Buffer solution (Placebo Comparator): Placebo solution (PBS) will be administered daily in the form of 1 mL of PBS (phosphate buffered saline) by inhalation
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: TPI ASM8 — Administered with the I-Neb device from Respironics once daily by inhalation over 2 treatment periods of 14 days each
  Arms: No.1 ASM8 (oligonucleotide)
Biological: placebo — Administered with the I-Neb device from Respironics once daily by inhalation over 2 treatment periods of 14 days each
  Arms: Phosphate Buffer solution

SUMMARY:
The researchers propose to study the airways of asthmatics given TPI ASM8 for 14 days, and examine the protective effects on allergen-induced bronchoconstriction, hyperresponsiveness and airway inflammation.

DETAILED DESCRIPTION:
Early and late asthmatic responses were attenuated by ASM8 and by placebo solution.Methacholine challenge was not affected by study medication. Other parameters were unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age
* Intermittent mild to moderate allergic asthma as defined by ATS/ERS criteria
* History of episodic wheeze and shortness of breath

Exclusion Criteria:

* Significant acute or chronic medical, neurologic, cardiovascular or psychiatric illness, asthma exacerbation or respiratory infection in the preceding 6 weeks
* Use of oral/injectable corticosteroids within the last 60 days or currently on any anti-asthmatic drugs, immunosuppressives, nonsteroidal anti-inflammatory drugs or anticoagulants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety and allergen-induced maximum decrease in FEV1 for Late Asthmatic Response | Safety (Trial duration) + LAR (Day 14)

SECONDARY OUTCOMES:
Exploratory Endpoints only: EAR on Day 14, AMP-induced airway hyperresponsiveness on Day 10,eNO on Day 14, PK/PD in sputum and plasma | study duration

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Connor, MD, Principal Investigator — Kings College Hospital, London, United Kingdom; Rene Pageau, M.Sc.Pharm, Study Director — Topigen Pharmaceuticals, Montreal, Quebec/Canada; Pierluigi Paggiaro, Prof, Principal Investigator — University of Pisa, Pisa, Italy; Dave Singh, MD, Principal Investigator — Evaluation Unit, Manchester, UK; Peter J. Sterk, MD, Principal Investigator — University of Amsterdam, Amsterdam, The Netherlands; Piero Maestrelli, Prof., Principal Investigator — University of Padova, Padova, Italy
Locations (1):
- King's College inLondon, London, London, United Kingdom